CLINICAL TRIAL: NCT00853918
Title: Clinical Practice Intensity: Comparing VA to Private Sector Providers
Brief Title: Clinical Practice Intensity: Comparing Veterans Affairs (VA) to Private Sector Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 03-242; DMS-17632 (Other Grant/Funding Number: White River Junction VAMC)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Physician Survey Response Rates
Keywords: Physician survey; Mail survey; Response rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- $20 Cash (Experimental)
  Interventions: Other: $20 cash
- $50 Cash (Experimental)
  Interventions: Other: $50 cash
- $50 Check (Experimental)
  Interventions: Other: $50 check
- $100 Check (Experimental)
  Interventions: Other: $100 check

INTERVENTIONS:
Other: $20 cash — $20 cash incentive mailed with survey
  Arms: $20 Cash
Other: $50 cash — $50 cash incentive mailed with survey
  Arms: $50 Cash
Other: $50 check — $50 check incentive mailed with survey
  Arms: $50 Check
Other: $100 check — $100 check incentive mailed with survey
  Arms: $100 Check

SUMMARY:
This is a national physician mail survey examining primary care practice patterns. The experimental component of the study (the clinical trial) is a randomized trial of different monetary incentive forms and amounts for physicians invited to participate in the study. Only non-VA physicians will be included in this part of the study. (VA physicians are not allowed to receive monetary incentives.) Physicians will be randomized to receive one of four incentives. The main outcome measure is the response rate.

DETAILED DESCRIPTION:
This primary care physician survey is being conducted by Harris Interactive, an international survey research firm working collaboratively under contract to VA investigators heading the study. Surveys will be mailed to a random sample of 1000 non-VA primary care general internists practicing 20 or more clinical hours per week, identified via the Physician Masterfile of the American Medical Association.

The initial survey mailing, delivered via USPS Priority Mail, will include a cover letter inviting the physician to participate, a 12-page survey booklet (including a cover page, a 9-page survey, and 2 blank pages), a monetary incentive, and a prepaid addressed return envelope. The survey is estimated to take 20 minutes to complete. All survey recipients will also have the opportunity, as part of the survey, to request information about practice patterns in their community. Harris Interactive will randomly assign all invited (non-VA) physicians to receive one of four incentives, included in the initial survey mailing.

Non-responders will be contacted two additional times (at approximately 2 and 4 weeks following the initial mailing) by telephone and by mail. Subsequent mailings will include the survey, a cover letter, and a stamped addressed return envelope, but no monetary incentive.

Response rates will be compared between the four arms of the trial; between check v. cash; and between different denominations.

ELIGIBILITY:
Inclusion Criteria:

* Primary care general internists in the United States, identified through the AMA Physician Masterfile, who practice at least 20 hours per week are eligible to participate.
* All physicians included in the sample to whom the survey packets are mailed will be included in the analysis of the incentive experiment, except those for whom a survey packet is returned as undeliverable and those non-respondents identified through follow-up procedures as non-locatable, deceased, or retired.

Exclusion Criteria:

- Physicians self-identified in the AMA Masterfile as medical subspecialists or hospitalists are excluded from the sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
Survey response rate | 2 weeks, 2 months (primary), and 6 months after initial mailing

SECONDARY OUTCOMES:
Item non-response rates | 2 weeks, 2 months (primary), and 6 months after initial mailing

CONTACTS AND LOCATIONS:
Overall Officials: Brenda E Sirovich, MD MS, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT

REFERENCES:
- [Result] Sirovich BE, Gottlieb DJ, Welch HG, Fisher ES. Regional variations in health care intensity and physician perceptions of quality of care. Ann Intern Med. 2006 May 2;144(9):641-9. doi: 10.7326/0003-4819-144-9-200605020-00007. PMID 16670133
- [Result] Robertson DJ, Sirovich BE. Colorectal cancer risk following a negative colonoscopy. JAMA. 2006 Nov 22;296(20):2437; author reply 2437-8. doi: 10.1001/jama.296.20.2437-a. No abstract available. PMID 17119136
- [Derived] Sirovich BE, Woloshin S, Schwartz LM. Too Little? Too Much? Primary care physicians' views on US health care: a brief report. Arch Intern Med. 2011 Sep 26;171(17):1582-5. doi: 10.1001/archinternmed.2011.437. PMID 21949169